CLINICAL TRIAL: NCT06675539
Title: Validation of the French Version of the Prediction of the Alcohol Withdrawal Severity Scale (PAWSS)
Acronym: PAWSS-VF
Status: Recruiting | Type: Observational
Sponsor: Etablissement Public de Santé Barthélemy Durand (Other)
Responsible Party: Sponsor
Other Study IDs: 24P04; 2022-A01364-39 (Registry Identifier: ANSM)
Record Dates: First submitted 2024-09-30; First posted 2024-11-05 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Addiction, Substance; Alcohol Use Disorder; Alcohol Dependence; Alcohol Withdrawal
Keywords: Alcohol Use Disorder; Scale; alcohol withdrawal; prediction; withdrawal syndrome
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism; Substance Withdrawal Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- AUD participant: Subject evaluation included during 3 days.
  Day 1: Collection of consent and clinical data, DSM-5 criterion for alcohol use disorders, AUDIT, PRSAC scale (twice by two investigators), and CIWA-AR scale every 8 hours.
  Day 2 and Day 3: administration of CIWA-AR scale every 8 hours.
  Interventions: Diagnostic Test: French version PAWSS

INTERVENTIONS:
Diagnostic Test: French version PAWSS — French version of the Prediction of Alcohol Withdrawal Severity Scale

SUMMARY:
The goal of this observational study is to validate the French version of the PAWSS scale in a population of patients with Alcohol Use Disorders. Prediction of Alcohol Withdrawal Severity Scale (PAWSS) has an excellent psychometric characteristics and predictive value of complicated alcohol withdrawal.

The main question it aims to answer is:

Are the psychometric properties of the French version of the PAWSS scale comparable to those of the English version in a population of alcohol use disorders subjects?

AUDs participants are included and followed for three days during their hospitalization, They will performed several scales and surveys (DSM-5 AUD criteria, AUDIT, French version of PAWSS and CIWA-AR).

DETAILED DESCRIPTION:
Context Alcohol use disorders (AUDs) are reported in 10-32% of hospitalized medical patients [Nielsen et al. 1994; Smothers et al. 2004; Dolman and Hawkes 2005; Doering-Silveira et al. 2014], in 23 % of hospitalized medical patients and in 25-50% of hospitalized psychiatric patients in France [Paille & Reynaud 2015]. A hospital admission may result in an abrupt cessation of alcohol consumption for individuals with AUD and thus provide a risk period for alcohol withdrawal syndrome. Even though the majority of patients at risk of AWS will develop only minor or uncomplicated withdrawal symptoms, up to 20% of patients develop symptoms associated with complicated alcohol withdrawal, including withdrawal seizures and delirium tremens [Maldonado et al., 2010]. Complicated alcohol withdrawal syndrome is associated with increased in-hospital morbidity and mortality, increased lengths of stay, inflated costs of care, and worsened cognitive functioning.

Due to lack of any similar previously existing tools, Maldonado et al. developed the Prediction of Alcohol Withdrawal Severity Scale (PAWSS) [Maldonado et al. 2014, 2015]. The PAWSS scale has excellent psychometric characteristics and predictive value of complicated alcohol withdrawal among medically ill hospitalized patients using a PAWSS cutoff of 4, the tool's sensitivity was 93.1% and specificity was 99.5%. The PAWSS scale is recommended by the American Society of Addiction Medicine for alcohol withdrawal management, (ASAM 2020, www.asam.org).

There is no scale available to identify the patients at risk of complicated withdrawal In France. The PAWSS is not a withdrawal severity scale such as the CIWA-AR or Cushman scale, which are scored during withdrawal, but a scale designed to screen beforehand, prior to withdrawal, patients at high risk for the most severe complications (Delirium tremens and seizures), and thus to take appropriate therapeutic measures. It also has the advantage of being able to guide patients towards the most suitable scheduled withdrawal modalities for their condition.

The PAWSS can therefore greatly assist clinicians in directing patients to either outpatient or hospital withdrawal in more or less intensive care, with a minimum of risk. Its use would allow earlier management to limit the sequelae, especially cognitive and those related to seizures.

The PAWSS scale includes an initial screener question and can be used with patients who are not currently exhibiting signs of withdrawal. If a patient does indeed endorse recent intake of alcohol, this must be followed by 10 questions contained in the second part of PAWSS, assessing known risk factors for withdrawal and current clinical status. The PAWSS is heavily based on self-report of alcohol intake and history provided by patients, as the literature suggests that interviews by clinicians can provide the most accurate information on alcohol abuse and relapse, as compared to collateral information or selected laboratory data.

Objectives The primary objective is to validate the French version of the PAWSS scale (PRSAC) in a population of patients with AUD.

The secondary objectives are 1) to confirm the optimal cut-off score of 4 for the PRSAC scale, 2) to evaluate PRSAC scale reproducibility in predicting the risk of complicated alcohol withdrawal syndrome and 3) to identify an optimal strategy for benzodiazepine use following the application of PRSAC scale.

Hypothesis Are the psychometric properties of the French version of the PAWSS scale (PRSAC) comparable to those of the English version in a population of alcohol use disorders subjects?

Methods This study is a multicentric non-interventional prospective cohort study. Subject evaluation included during 3 days.

Day 1: Collection of consent and clinical data, DSM-5 criterion for alcohol use disorders, AUDIT, PRSAC scale (twice by two investigators), and CIWA-AR scale every 8 hours.

Day 2 and Day 3: administration of CIWA-AR scale every 8 hours.

Inclusion criteria Male or female, aged 18 to 60 years Subjects with DSM-5 criteria for moderate to severe alcohol use disorders (AUD) Subjects hospitalized for AUD or another condition with AUD. Subjects who understand French and affiliated to the social security system

Non-inclusion criteria Subject with a neurological disorder, impairing cognition (epilepsy, dementia,…) Subjects unable to understand the questionnaire and to give consent or not volunteering for the study Subject under guardianship or curatorship

Study location

Academic substance abuse treatment and Psychiatry departments of:

Barthélemy Durand Hospital at Etampes, France Paul Brousse hospital in Villejuif, France Rouen university hospital, France Caen university hospital, France Martinique university hospital, France

Results & Outcome Confirmation of the psychometric qualities of the French version of the PAWSS scale.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 60 years
* Subjects with DSM-5 criteria for alcohol use disorders (AUD)
* Subjects hospitalized for scheduled withdrawal or patients developing alcohol withdrawal hospitalized for another reason.
* Subjects who understand French
* Subject affiliated to the French social security system
* Subject having given their written consent to the study

Exclusion Criteria:

* Subjects transferred from other hospitalization services for whom a withdrawal syndrome could have already been treated.
* Subjects scheduled for discharge within 48 hours.
* Subjects with known uncontrolled epilepsy.
* Subjects unable to understand the questionnaire.
* Subjects unable to give consent or not volunteering for the study.
* Subjects under guardianship or curatorship.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: AUD adults subjects hospitalized
Sampling Method: Non-Probability Sample
Enrollment: 545 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Psychometric qualities evaluation of French PAWSS | 3 days
  The primary endpoint is the evaluation of the psychometric qualities of the French version of PAWSS scale (PRSAC) by measuring predictive performance through the calculation of sensitivity, specificity, and positive and negative predictive values.

SECONDARY OUTCOMES:
The optimal cut-off score of 4 for the French version of the Prediction of the Alcohol Withdrawal Severity Scale | 3 days
  The optimal cut-off score of 4 will be determined by ROC curve analysis to confirm the cut-off for the French version of the Prediction of Alcohol Withdrawal Severity Scale. A French version of the Prediction of the Alcohol Withdrawal Severity Scale score of 4 or higher indicates a high risk of developing a complicated withdrawal syndrome.
Reproducibility in predicting the risk of French PAWSS | 3 days
  Evaluate the reproducibility of the French version of the Prediction of the Alcohol Withdrawal Severity Scale in predicting the risk of complicated alcohol withdrawal syndrome by measuring inter-rater reliability through the calculation of Cohen's Kappa and Lin's concordance coefficients.
Doses and Durations of Benzodiazepine | 3 days
  The doses and durations of benzodiazepine use during the study are collected during each participant's involvement in the study. These doses and durations will be compared between a group with a score below 4 and a group with a score of 4 or higher on the French version of the Prediction of Alcohol Withdrawal Severity Scale

CONTACTS AND LOCATIONS:
Overall Officials: Alain Dervaux, Principal Investigator — Etablissement Public de Santé Barthélemy Durand
Locations (1):
- Etablissement Public de Santé Barthélemy Durand, Étampes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maldonado JR, Sher Y, Das S, Hills-Evans K, Frenklach A, Lolak S, Talley R, Neri E. Prospective Validation Study of the Prediction of Alcohol Withdrawal Severity Scale (PAWSS) in Medically Ill Inpatients: A New Scale for the Prediction of Complicated Alcohol Withdrawal Syndrome. Alcohol Alcohol. 2015 Sep;50(5):509-18. doi: 10.1093/alcalc/agv043. Epub 2015 May 21. PMID 25999438
- [Background] Maldonado JR, Sher Y, Ashouri JF, Hills-Evans K, Swendsen H, Lolak S, Miller AC. The "Prediction of Alcohol Withdrawal Severity Scale" (PAWSS): systematic literature review and pilot study of a new scale for the prediction of complicated alcohol withdrawal syndrome. Alcohol. 2014 Jun;48(4):375-90. doi: 10.1016/j.alcohol.2014.01.004. Epub 2014 Feb 19. PMID 24657098
- [Background] Campos J, Roca L, Gude F, Gonzalez-Quintela A. Long-term mortality of patients admitted to the hospital with alcohol withdrawal syndrome. Alcohol Clin Exp Res. 2011 Jun;35(6):1180-6. doi: 10.1111/j.1530-0277.2011.01451.x. Epub 2011 Feb 25. PMID 21352245
- [Background] Eloma AS, Tucciarone JM, Hayes EM, Bronson BD. Evaluation of the appropriate use of a CIWA-Ar alcohol withdrawal protocol in the general hospital setting. Am J Drug Alcohol Abuse. 2018;44(4):418-425. doi: 10.1080/00952990.2017.1362418. Epub 2017 Oct 5. PMID 28981333
- [Background] Sullivan JT, Sykora K, Schneiderman J, Naranjo CA, Sellers EM. Assessment of alcohol withdrawal: the revised clinical institute withdrawal assessment for alcohol scale (CIWA-Ar). Br J Addict. 1989 Nov;84(11):1353-7. doi: 10.1111/j.1360-0443.1989.tb00737.x. PMID 2597811